CLINICAL TRIAL: NCT05216809
Title: The Efficacy of a Non-Invasive 13CO2 'Breath Test' to Detect Anabolic Resistance Following Step Reduction in Younger and Older Adults
Brief Title: Oral 'Breath Test' to Measure Anabolic Sensitivity in Young and Older Adults at Different Activity Levels
Acronym: ARBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Principal Investigator, University of Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ARBT
Record Dates: First submitted 2021-11-07; First posted 2022-02-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Sedentary Behavior; Aging; Sarcopenia; Amino Acids; Dietary Protein
Keywords: Skeletal Muscle; Step-Reduction; Aging; Anabolic Resistance; Physical Activity; Stable Isotopes
MeSH Terms: conditions — Sedentary Behavior; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Group Cohort Study
  Twenty healthy young (18-35 years of age; 10 females and 10 males) and twelve healthy older adults (60-80 years of age; 6 females and 6 males), for a total of 32 individuals, will undergo 3 days (Days 1-3) of Habitual Activity in a free-living setting (Phase 1) followed by a metabolic trial (Day 4), where individuals will be subjected to a non-invasive 13CO2 breath-test. This will also serve as a lead-in period for the subsequent 3 days of step-reduction (<2,000 steps/day; Days 4-6). Following the 3-days of reduced daily step count (Day 7), participants will undergo another metabolic trial day involving the non-invasive 13CO2 breath-test in order for us to determine changes in anabolic sensitivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Adults (Active Comparator): Equal sex distribution (10M/10F); ages 18-35 years old.
  Interventions: Behavioral: Habitual Physical Activity; Behavioral: Step-Reduction
- Older Adults (Active Comparator): Equal sex distribution (6M/6F); ages 60-80 years old.
  Interventions: Behavioral: Habitual Physical Activity; Behavioral: Step-Reduction

INTERVENTIONS:
Behavioral: Habitual Physical Activity — Participants will maintain habitual levels of physical activity (inclusive of structured physical activity). Participants will be required to maintain >7,000 steps/day.
  Other Names: Free-Living Activity
Behavioral: Step-Reduction — Participants will be required to reduce their daily step-counts to <2,000 steps/day. Further, they will be required to refrain from structured physical activity.
  Other Names: Reduced Physical Activity

SUMMARY:
Recent work in the investigators laboratory has examined the ability of a non-invasive 13CO2 breath-test to assess differences in amino acid oxidation rates and net balance in young healthy males following protein feeding and resistance exercise. The investigators aim to test the efficacy of this non-invasive 13CO2 breath-test to assess for differences in anabolic sensitivity between young and older adults following an acute period of habitual and reduced physical activity.

DETAILED DESCRIPTION:
Aging is associated with a phenomenon known as anabolic resistance, whereby individuals are less responsive to anabolic stimuli (i.e., resistance exercise, dietary protein ingestion). Mild and severe reductions in physical activity are also known to play a key role in the emergence of anabolic resistance. Therefore, the purpose of this study is to investigate the ability of a non-invasive 13CO2 breath-test to assess differences in whole-body leucine oxidation and leucine net balance between younger and older individuals under conditions of habitual activity and following a period of reduced activity/step-reduction. In this manner, the ability of the methodology to distinguish anabolic sensitivity between young and older adult populations will be assessed.

Methods:

Total participant time commitment will span over 4 sessional dates:

Session 1 - Introduction Interested participants will be recruited to engage in a video conference call to undergo an introductory session. Participants will be provided with a comprehensive introduction to the study which will explain the research objectives, conduct, and associated risks. Participants will provide informed consent prior to the collection of any study information (i.e., anthropometrics and habitual activity levels). Eligibility will also be screened for at this time.

Session 2 - Body Composition Assessment Participants will consume a bolus of deuterium oxide (D2O) and provide saliva samples in order to estimate fat-free mass.

The remainder of the study will consist of seven consecutive days, wherein Phase 1 (Habitual Activity) will be subsequently followed by Phase 2 (Step-Reduction).

Phase 1 - Habitual Activity (Days 1-3) Participants will be asked to engage in their habitual activity pattern (> 7000 steps/day) while wearing an accelerometer and pedometer. Participants will be further instructed to maintain their normal dietary patterns and to track their diets over the course of these three days using diet logs.

Session 3 - Habitual Activity Metabolic Trial (Day 4) On the morning of the fourth day, following three days of habitual activity, participants will be subjected to the non-invasive 13CO2 breath-test to assess for whole-body leucine oxidation and net balance. This date will also serve as a lead-in to the subsequent Phase 2.

Phase 2 - Step-Reduction (Days 4-6) Participants will be asked to maintain their normal dietary patterns and track their dietary intake, but will need to adhere to a reduced daily step count (<2000 steps/day). Accelerometers and pedometers will be worn again during this period.

Session 4 - Step-Reduction Metabolic Trial (Day 7) On the morning of the 7th day, following three days of reduced daily step-count, participants will be subjected again to the non-invasive 13CO2 breath-test to assess for whole-body leucine oxidation and net balance. Ultimately, this will allow us to determine whether 3-days of reduced step-count will impart any changes on anabolic sensitivity.

For each metabolic trial, two urine samples (baseline and pooled enriched) will be collected, in addition to breath samples collected over a 6-hour post-prandial period at 20-30 minute intervals. These biological samples will be used to measure tracer excretion and oxidation, allowing us to determine rates of protein metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young (age: 18-35 years) or older (age: 60-80 years) adults
* Average daily step-count >7,000/day
* BMI between normal to overweight (18.5-29.9 kg/m2)

Exclusion Criteria:

* Regular use of nonsteroidal anti-inflammatory drugs (with the exception of daily low-dose aspirin)
* Use of anticoagulants
* Use of a walker, cane, or assistive walking device
* Current or recently remised cancer
* Infectious or gastrointestinal disease
* Inability to comply with study protocol (e.g., >2,000 steps/day during Step-Reduction Phase)
* Regular tobacco use
* Self-reported illicit drug use (e.g. growth hormone, testosterone, etc.)
* Diagnosed chronic illness (e.g. type 2 diabetes, heart disease, thyroid disease)
* Pregnant
* Hormonal Replacement Therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Exogenous Leucine Oxidation (umol/kg) | 6 hours
  Exogenous Leucine Oxidation determined from breath 13CCO2 enrichment. Breath samples will be collected every 20-30min after test drink ingestion to determine breath 13CO2 enrichment. Total leucine oxidation will be determined from the area under the 13CO2 enrichment by time curve.
Net Leucine Retention (umol/kg) | 6 hours
  Whole-Body Net Leucine Retention determined from the difference between exogenous leucine oxidation and leucine ingestion the 6 hour measurement period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, PhD, Principal Investigator — University of Toronto; Hugo JW Fung, PhD (c), Study Director — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No